CLINICAL TRIAL: NCT02980653
Title: A Phase II Study Assessing the Efficacy of Prophylaxis Use of Megestrol Acetate Against Cancer-related Critical Body Weight Loss in Patients With Head and Neck Cancer Who Receiving Concurrent Chemoradiotherapy
Brief Title: Megestrol Acetate Against Cancer-related Critical Body Weight Loss in Patients With H&N Cancer Who Receiving CCRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TTY Biopharm (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TTYMG1403
Record Dates: First submitted 2016-07-25; First posted 2016-12-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Head and Neck Cancer
Keywords: Phase II study; Critical body weight loss; Concurrent chemoradiotherapy; Megestrol acetate; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Megestrol (Experimental): Single arm
  Interventions: Drug: Megestrol acetate (MA) 400 mg/day

INTERVENTIONS:
Drug: Megestrol acetate (MA) 400 mg/day — Megestrol acetate (MA) will be given on 400 mg/day as eligible patient begin CCRT. Total treatment period is for a maximum of 12 weeks calculated from the date of first dose.
  Other Names: Megest

SUMMARY:
Primary Objective:

To evaluate the population prevalence of critical body weight loss ( more than 5% from baseline) in patients with Head and Neck cancer.

Secondary Objectives:

To evaluate the impact of appetite, and performance status; To evaluate the change of quality of life (QoL); To evaluate the incidence of infection and hospitalization; To evaluate the safety profiles

DETAILED DESCRIPTION:
Hypothesis testing will be used to determine the patient number in this study. According to a preliminary data at CGMH-LK, the investigators have the untreated patients with population prevalence of critical weight loss that is 0.56, and the investigators assume the study treated population prevalence is 0.4, power set in 0.9, alpha set in 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is confirmed the diagnosis of head and neck cancer and will receive concurrent chemoradiotherapy (CCRT).
* Patient who is capable to understand and complete questionnaires
* Patient who is convenient to receive body weight measurement
* Life expectancy of at least 12 weeks
* Age over 20 years old at registration
* Voluntarily signed the written informed consent form

Exclusion Criteria:

* Special populations that needs unique risk/benefit considerations. (Ex. Pregnant or nursing women or mental disorder patients, et al.)
* Any significant co-morbid medical condition that out of medication control. (Ex. Heart/renal/hepatic failure or poorly controlled diabetes, et al.)
* Any evidence of mechanical obstruction of the alimentary track, malabsorption, or intractable vomiting.
* Any thromboembolism event, e.g. cerebral or peripheral vascular disease
* Judged ineligible by physicians for participation in the study due to any safety concern.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Critical body weight loss | 12 weeks
  To evaluate the population prevalence of critical body weight loss ( > 5% from baseline) in patients with Head and Neck cancer

SECONDARY OUTCOMES:
Impact of appetite | 12 weeks
  The assessment of appetite will be performed before the entry of the study, and then repeated every visit until end of study. The assessment of appetite will be performed by the visual analogue scale(VAS) within the range of 0-100mm(please refer Appendix II). The Differences from baseline status will be assessed, and results will be presented in percentages of improved patients out of those treated at the time of evaluation.
Impact of performance status | 12 weeks
  The assessment of appetite will be performed before the entry of the study, and then repeated every visit until end of study. The measurement will base on ECOG performance status scale(please refer Appendix I). The Differences from baseline status will be assessed, and results will be presented in percentages of improved patients out of those treated at the time of evaluation.
Change of quality of life (QoL) | 12 weeks
  Quality of life (QOL) will be evaluated since patient registration to off study by means of the Functional Assessment of Cancer Therapy-Head and Neck (FACT-. H&N), Version 4 (Traditional Chinese) (please refer Appendix III). The questionnaire will be completed under the assistance of a trained study nurse.
Incidence of infection and hospitalization | 12 weeks
  If any patient in the study period (3 months) suffer infection or hospitalization, that should be recorded on Case Report Form for the descriptive statistics analysis.
Safety profiles (percentage of patients with at least one occurrence of preferred term will be included, according to the most severe NCI-CTCAE v4.03 grade) | 12 weeks
  Adverse event / toxicity assessment are based on NCI- Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03), please refer Appendix IV), and will be evaluated before the treatment, and then repeated each visit until off study. The incidence and percentage of patients with at least one occurrence of preferred term will be included, according to the most severe NCI-CTCAE v4.03 grade.

OTHER OUTCOMES:
Measurability of Anthropometric Evaluation | 12 weeks
  Anthropometric evaluation is including body weight and body mass index.
Lab test | 12 weeks
  Lab test should be conducted every patient's visit for safety assessment. CRP and TNFα will be exanimated at screening and every 4 weeks of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Ming Wang, M.D., Principal Investigator — Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (1):
- Chang-Gung Memorial Hospital, Linkou, Linkou District, Taiwan

REFERENCES:
- [Background] Kumar NB, Kazi A, Smith T, Crocker T, Yu D, Reich RR, Reddy K, Hastings S, Exterman M, Balducci L, Dalton K, Bepler G. Cancer cachexia: traditional therapies and novel molecular mechanism-based approaches to treatment. Curr Treat Options Oncol. 2010 Dec;11(3-4):107-17. doi: 10.1007/s11864-010-0127-z. PMID 21128029
- [Background] Vadell C, Segui MA, Gimenez-Arnau JM, Morales S, Cirera L, Bestit I, Batiste E, Blanco R, Jolis L, Boleda M, Anton I. Anticachectic efficacy of megestrol acetate at different doses and versus placebo in patients with neoplastic cachexia. Am J Clin Oncol. 1998 Aug;21(4):347-51. doi: 10.1097/00000421-199808000-00006. PMID 9708631
- [Background] Pascual Lopez A, Roque i Figuls M, Urrutia Cuchi G, Berenstein EG, Almenar Pasies B, Balcells Alegre M, Herdman M. Systematic review of megestrol acetate in the treatment of anorexia-cachexia syndrome. J Pain Symptom Manage. 2004 Apr;27(4):360-9. doi: 10.1016/j.jpainsymman.2003.09.007. PMID 15050664
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Inui A. Cancer anorexia-cachexia syndrome: current issues in research and management. CA Cancer J Clin. 2002 Mar-Apr;52(2):72-91. doi: 10.3322/canjclin.52.2.72. PMID 11929007
- [Background] Maltoni M, Nanni O, Scarpi E, Rossi D, Serra P, Amadori D. High-dose progestins for the treatment of cancer anorexia-cachexia syndrome: a systematic review of randomised clinical trials. Ann Oncol. 2001 Mar;12(3):289-300. doi: 10.1023/a:1011156811739. PMID 11332139
- [Background] Beller E, Tattersall M, Lumley T, Levi J, Dalley D, Olver I, Page J, Abdi E, Wynne C, Friedlander M, Boadle D, Wheeler H, Margrie S, Simes RJ. Improved quality of life with megestrol acetate in patients with endocrine-insensitive advanced cancer: a randomised placebo-controlled trial. Australasian Megestrol Acetate Cooperative Study Group. Ann Oncol. 1997 Mar;8(3):277-83. doi: 10.1023/a:1008291825695. PMID 9137798
- [Background] De Conno F, Martini C, Zecca E, Balzarini A, Venturino P, Groff L, Caraceni A. Megestrol acetate for anorexia in patients with far-advanced cancer: a double-blind controlled clinical trial. Eur J Cancer. 1998 Oct;34(11):1705-9. doi: 10.1016/s0959-8049(98)00219-6. PMID 9893656
- [Background] Gebbia V, Testa A, Gebbia N. Prospective randomised trial of two dose levels of megestrol acetate in the management of anorexia-cachexia syndrome in patients with metastatic cancer. Br J Cancer. 1996 Jun;73(12):1576-80. doi: 10.1038/bjc.1996.297. PMID 8664133
- [Background] Loprinzi CL, Michalak JC, Schaid DJ, Mailliard JA, Athmann LM, Goldberg RM, Tschetter LK, Hatfield AK, Morton RF. Phase III evaluation of four doses of megestrol acetate as therapy for patients with cancer anorexia and/or cachexia. J Clin Oncol. 1993 Apr;11(4):762-7. doi: 10.1200/JCO.1993.11.4.762. PMID 8478668
- [Background] Tchekmedyian NS, Hickman M, Siau J, Greco FA, Keller J, Browder H, Aisner J. Megestrol acetate in cancer anorexia and weight loss. Cancer. 1992 Mar 1;69(5):1268-74. doi: 10.1002/cncr.2820690532. PMID 1739926
- [Background] Tomiska M, Tomiskova M, Salajka F, Adam Z, Vorlicek J. Palliative treatment of cancer anorexia with oral suspension of megestrol acetate. Neoplasma. 2003;50(3):227-33. PMID 12937858
- [Background] Rogers LQ, Rao K, Malone J, Kandula P, Ronen O, Markwell SJ, Courneya KS, Robbins KT. Factors associated with quality of life in outpatients with head and neck cancer 6 months after diagnosis. Head Neck. 2009 Sep;31(9):1207-14. doi: 10.1002/hed.21084. PMID 19360748
- [Background] McRackan TR, Watkins JM, Herrin AE, Garrett-Mayer EM, Sharma AK, Day TA, Gillespie MB. Effect of body mass index on chemoradiation outcomes in head and neck cancer. Laryngoscope. 2008 Jul;118(7):1180-5. doi: 10.1097/MLG.0b013e31816fca5c. PMID 18475213
- [Background] Couch ME, Dittus K, Toth MJ, Willis MS, Guttridge DC, George JR, Barnes CA, Gourin CG, Der-Torossian H. Cancer cachexia update in head and neck cancer: Definitions and diagnostic features. Head Neck. 2015 Apr;37(4):594-604. doi: 10.1002/hed.23599. Epub 2014 Mar 25. PMID 24415363
- [Background] Capuano G, Grosso A, Gentile PC, Battista M, Bianciardi F, Di Palma A, Pavese I, Satta F, Tosti M, Palladino A, Coiro G, Di Palma M. Influence of weight loss on outcomes in patients with head and neck cancer undergoing concomitant chemoradiotherapy. Head Neck. 2008 Apr;30(4):503-8. doi: 10.1002/hed.20737. PMID 18098310
- [Background] Mantovani G, Maccio A, Bianchi A, Curreli L, Ghiani M, Santona MC, Del Giacco GS. Megestrol acetate in neoplastic anorexia/cachexia: clinical evaluation and comparison with cytokine levels in patients with head and neck carcinoma treated with neoadjuvant chemotherapy. Int J Clin Lab Res. 1995;25(3):135-41. doi: 10.1007/BF02592554. PMID 8562975
- [Background] Donohoe CL, Ryan AM, Reynolds JV. Cancer cachexia: mechanisms and clinical implications. Gastroenterol Res Pract. 2011;2011:601434. doi: 10.1155/2011/601434. Epub 2011 Jun 13. PMID 21760776
- [Background] Capozzi LC, Lau H, Reimer RA, McNeely M, Giese-Davis J, Culos-Reed SN. Exercise and nutrition for head and neck cancer patients: a patient oriented, clinic-supported randomized controlled trial. BMC Cancer. 2012 Oct 2;12:446. doi: 10.1186/1471-2407-12-446. PMID 23031071